CLINICAL TRIAL: NCT04802824
Title: Determining the Magnitude of Change in [18F]FPIA-detectable Short Chain Fatty Acid Uptake in Metastatic Renal Cell Cancer Following Therapy
Brief Title: Measuring Treatment Response in Metastatic Renal Cell Cancer Using FPIA PET/CT
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20CX6143
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: PET/CT; Fatty Acid Oxidation
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival tumour biopsies from the primary or metastatic lesion, taken within 3 months of the first [18F]FPIA PET/CT scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PET/CT — 18F-fluoropivalate PET/CT scan.
  Other Names: Imaging Scan

SUMMARY:
Renal cell carcinoma (RCC) is the most prevalent and lethal malignancy of the kidney. At the time of diagnosis, as many as a fifth of patients have metastatic disease (mRCC). Despite advances in treatment, long-term survival rates remain poor. 18F-fluoropivalate ([18F]FPIA) is a new tracer that images short chain fatty acid (SCFA) uptake in tumours, a key component of fatty acid oxidation.

The aim of the study is to investigate longitudinal changes in [18F]FPIA uptake at baseline, at 4-6 weeks and at 12 weeks following treatment initiation in patients using tyrosine kinase inhibitors (TKI's), chemotherapy, immunotherapy, or combinations of these.

The investigators hypothesise that the import of [18F]FPIA-detectable SCFA into tumours is high and decreases with effective treatment.

DETAILED DESCRIPTION:
24 evaluable patients with radiological and/or histological evidence of mRCC and due to receive systemic therapy will be enrolled. The patients invited to participate in the study will provide written informed consent. Patients will only undergo [18F]FPIA positron emission tomography (PET)/computed tomography (CT) imaging once they have satisfied the inclusion and exclusion criteria. Once these have been satisfied, eligible patients will proceed to [18F]FPIA PET/CT. Patients will have three imaging visits at baseline, 4-6 weeks and 12 weeks post the commencement of treatment. Patients will have been treated as per standard of care, which may have included TKI's, chemotherapy, immunotherapy or combinations of these. Data will be considered complete when patients have all three analysable scans. In the event of dropout, additional subjects will be recruited to reach a total number of 24 evaluable subjects.

On each day of imaging the patients will have a blood test and a urine sample collected to measure concentrations of carnitine. For each scan, a single dose of [18F]FPIA (maximum 370 MBq) IV will be administered to the participant. The participant will then rest in a quiet place for an uptake period and undergo whole body PET/CT scanning from 60 minutes.

Archival tumour biopsies (primary or metastatic lesion), taken within 3 months of the 1st [18F]FPIA PET/CT scan will be retrieved for analysis where possible.

ELIGIBILITY:
Inclusion Criteria:

Patients with radiological and/or histological evidence of evidence of mRCC who are either:

A. Treatment naïve or newly relapsed (not currently on treatment)

or

B. Progressing on standard of care systemic therapy

and

C. That fulfil the following criteria:

1. Age ≥18
2. Target metastases size ≥ 1cm (outside of the liver).
3. The subject has an available diagnostic tumour biopsy of the primary and/or metastatic lesion taken within 3 months of the first [18F]FPIA PET/CT.
4. WHO performance status 0 - 2.
5. If female, the subject is either post-menopausal (>1 year), or surgically sterilized (has had a documented bilateral oophorectomy and/or documented hysterectomy, >2 years), or if of childbearing potential, must have a negative urine pregnancy test at initial screening and/or within 2 hours prior to injection of imaging agent.
6. eGFR of ≥30 within 3 months of [18F]FPIA injection
7. The subject is able and willing to comply with study procedures, and a signed and dated informed consent is obtained.
8. The subject is not scheduled to start cancer treatment prior to the first study PET/CT scan.

Exclusion Criteria:

1. Pregnant or lactating women
2. Evidence of significant medical condition or laboratory finding which, in the opinion of the Investigator, makes it undesirable for the patient to participate in the trial
3. The subject is receiving or has received chemotherapy, immunotherapy, biologic therapy or investigational therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of [18F]FPIA injection.
4. The subject is scheduled to have a nuclear medicine or contrast scan within 24 hours of the administration of [18F]FPIA.
5. Participants with claustrophobia or who are unable to comfortably tolerate the scanning procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiological and/or histological evidence of mRCC and due to receive systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Quantitative longitudinal measurement of [18F]FPIA uptake in mRCC. | Baseline, 4-6 weeks and 12 weeks post-commencement of treatment.
  PET/CT

SECONDARY OUTCOMES:
Quantitative measurement of FPIA in healthy tissue including kidneys. | Baseline, 4-6 weeks and 12 weeks post-commencement of treatment.
  PET/CT
Comparison of [18F]FPIA relative to baseline at 4-6 weeks and at 12 weeks (± 4 weeks) to changes on a patient's routine imaging scan. | Baseline, 4-6 weeks and 12 weeks post-commencement of treatment.
  Routine Imaging Scans - Determined by the NHS Treating Clinician.

OTHER OUTCOMES:
[18F]FPIA uptake versus Foundation Medicine mutational signature test (Tumour Mutational Burden (TMB)) on biopsy material. | Through study completion, an average of 3 years.
  Foundation Medicine mutational signature test.
[18F]FPIA uptake versus serum or urine carnitine/carnitine ester signature. | Through study completion, an average of 3 years.
  Serum and urine carnitine analysis at external laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust/Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT04802824/Prot_SAP_000.pdf